CLINICAL TRIAL: NCT03557203
Title: Dermatologic Tacrolimus Ointment on Eyelids in the Treatment of Steroid Refractory Vernal Keratoconjunctivitis and Atopic Keratoconjunctivitis
Brief Title: Dermatologic Tacrolimus Ointment on Eyelids in the Treatment of Refractory Vernal Keratoconjunctivitis and Atopic Keratoconjunctivitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201804062RIND
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-05

CONDITIONS: Vernal Keratoconjunctivitis; Atopic Keratoconjunctivitis; Tacrolimus
Keywords: Vernal Keratoconjunctivitis; Atopic Keratoconjunctivitis; tacrolimus
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the therapeutic effects of dermatologic tacrolimus ointment on eyelids to treat refractory vernal keratoconjunctivitis and atopic keratoconjunctivitis.

DETAILED DESCRIPTION:
Treatment of vernal keratoconjunctivitis (VKC) and atopic keratoconjunctivitis (AKC) is a challenge for the ophthalmologist and patients because of its wide variation in presentation and recurrence in nature. Patients has to be dependent on long term steroid control and suffered from complications, such as steroid glaucoma and secondary infection. About 32% of VKC patients is refractory to steroid treatment and another 35.4% of patients showed partial response. Tacrolimus ointment or eye drops are promising anti-inflammatory agents that have been shown very effective against VKC for patients suffering from severe VKC resistant to topical cyclosporine. Although tacrolimus eye drops is very effective in severe cases of VKC, unfortunately, it is only available in limited countries. Because of the unavailability of tacrolimus eye drops and side effect of long-tern steroid use, we tried to find other options for these severe VKC and AKC. Because there will be concomitant atopic dermatitis in the eyelid of severe cases of VKC and AKC, we retrospectively collected in cases using topical tacrolimus dermatological ointment on the skin of upper eye lid in the treatment of severe VKC and AKC with concomitant atopic dermatitis. Here, we reported 10 cases with either VKC or AKC whose symptoms resolved significantly with dermatologic tacrolimus ointment applying on eyelids.

ELIGIBILITY:
Inclusion Criteria:

* all patients diagnosed as severe vernal keratoconjunctivitis or atopic Keratoconjunctivitis and received topical dermatological tacrolimus ointment on upper eyelids between January, 2016 and January, 2018 at National Taiwan University Hospital.

Exclusion Criteria:

* none

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Severe vernal keratoconjunctivitis or atopic Keratoconjunctivitis diagnosed at the National Taiwan University Hospital (NTUH)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
serial external ocular photography and full chart records of patients who diagnosed as patients diagnosed as severe vernal keratoconjunctivitis and atopic keratoconjunctivitis refractory to steroid treatment | 2018/6/1-2019/5/31
  A retrospective review of charts and external ocular photography of all patients diagnosed as severe VKC or AKC and received topical dermatological tacrolimus ointment on upper eyelids between January, 2016 and January, 2018 at National Taiwan University Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: I-Jong Wang, professor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan